CLINICAL TRIAL: NCT07005336
Title: A Phase II, Randomized, Multicenter, Open-Label Study to Compare Uliledlimab Combined With Sintilimab and Chemotherapy Versus Sintilimab Combined With Chemotherapy in Patients With Previously Untreated Locally Advanced Unresectable or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study to Compare Uliledlimab Combined With Sintilimab and Chemotherapy Versus Sintilimab Combined With Chemotherapy in Patients With Previously Untreated Locally Advanced Unresectable or Metastatic Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ004309LUC201
Record Dates: First submitted 2025-05-21; First posted 2025-06-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Pemetrexed; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Non-squamous
  Squamous
  Interventions: Drug: Uliledlimab; Drug: Sintilimab; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Cisplatin Or Carboplatin
- Group B (Experimental): Non-squamous
  Squamous
  Interventions: Drug: Sintilimab; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Cisplatin Or Carboplatin

INTERVENTIONS:
Drug: Uliledlimab — 30 mg/kg, administered on Days 1 and 8 of Cycle 1 (C1D1 and C1D8), then once every 3 weeks (Q3W) starting from C2D1,at most 35 cycles
  Arms: Group A
Drug: Sintilimab — Intravenous infusion at a recommended dose of 200 mg once every 3 weeks，at most 35 cycles
Drug: Pemetrexed — Intravenously at a recommended dose of 500 mg/m2 body surface area (BSA) ,once every 3 weeks until the disease progresses.
Drug: Gemcitabine — 1000 mg/m2, administered on Days 1 and 8 ,once every 3 weeks (Q3W) for 4 cycles
Drug: Cisplatin Or Carboplatin — Cisplatin: 5 mg/m2 administered intravenously every 3-4 weeks for 4 cycles
  Carboplatin:75 mg/m2, administered intravenously every 3-4 weeks for 4 cycles

SUMMARY:
This is a Phase II, randomized, open-label, active-controlled, multicenter study to compare intravenous uliledlimab combined with sintilimab and chemotherapy versus sintilimab combined with chemotherapy in patients with previously untreated locally advanced unresectable or metastatic NSCLC who are not suitable for targeted therapies such as EGFR or ALK.

Eligible subjects will be randomly assigned in a 1:1 ratio to receive either uliledlimab combined with sintilimab and chemotherapy or sintilimab combined with chemotherapy. Enrolled subjects will first enter a safety run-in period. When at least 12 subjects have been randomly assigned to Group A and have received ≥ 1 dose of study drug (with a total of approximately 24 subjects), enrollment will be suspended for safety evaluation. The safety evaluation period will last 3 weeks, during which safety, tolerability, and PK data of uliledlimab combined with sintilimab and chemotherapy will be collected and evaluated by the Safety Review Committee (SRC). The SRC will decide through discussion whether to proceed to the next stage of randomized enrollment, whether additional subjects need to be enrolled for safety evaluation, or whether the study treatment should be terminated due to high safety risks. After the SRC reaches a unanimous resolution, enrollment will continue until a total of approximately 150 subjects are enrolled. All 150 subjects will be included in the final efficacy analysis. If 3 or more subjects experience Grade ≥ 3 treatment-related AEs that are unrelieved and lead to discontinuation of all study drugs during the safety run-in period, enrollment in the next stage will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years at the time of signing the ICF.
2. Patients with histologically or cytologically confirmed stage IIIB, IIIC, or IV NSCLC who are not suitable for radical surgery and/or radiotherapy.
3. Patients who have not received prior systemic therapy for their locally advanced or metastatic diseases.
4. Patients with measurable lesions as assessed by the investigator at the study site based on RECIST v1.1. Target lesions located in a previously irradiated region will be considered measurable only if there is documented evidence of disease progression.
5. Patients with non-squamous NSCLC who are confirmed to have no EGFR-sensitive mutations or ALK fusions.
6. atients with known PD-L1 and CD73 expression status in tumor tissue: it will be tested by the central laboratory for PD-L1 expression levels using the PD-L1 IHC 22C3 pharmDx assay, and CD73 expression levels using the CD73 antibody assay.
7. Patients with a life expectancy of at least 3 months.
8. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Patients with adequate organ function.
10. Patients with negative HIV testing at screening.
11. Patients with negative hepatitis B virus surface antigen (HBsAg) or inactive hepatitis B (HBsAg positive with HBV-DNA copy number ≤ ULN, ALT ≤ ULN, and no treatment is required in the investigator's opinion) at screening.
12. Patients with negative hepatitis C virus (HCV) antibody at screening, or positive HCV antibody and negative HCV RNA at screening.
13. For women of childbearing potential:A urine or serum pregnancy test must be negative within 72 hours prior to the first dose of study drug. If the urine pregnancy test result is positive or cannot be confirmed as negative, a serum pregnancy test should be performed.
14. For male subjects with female partners of childbearing potential:They must agree to use an effective method of contraception from the first dose of study drug to 180 days after the last dose of study drug.Male subjects with pregnant partners will be required to agree to use condoms; pregnant partners will not be required to use additional methods of contraception.
15. Patients who voluntarily agree to participate in the study and sign a written ICF.

Exclusion Criteria:

1. Patients who are currently pregnant, breastfeeding, or planning to conceive or give birth within the expected duration of this study.
2. Patients previously treated with immune checkpoint inhibitors or CD73 inhibitors.
3. Patients who are receiving or have completed systemic immune agonist therapy (including but not limited to: interferon, interleukin-2, and thymosin) within 4 weeks prior to the first dose or 5 drug elimination half-lives (whichever is longer).
4. Patients who have received oral or intravenous antibiotic therapy within 2 weeks prior to starting study treatment, except for prophylactic use.
5. Patients who have undergone major surgery within 4 weeks prior to starting study treatment, except for diagnostic surgery.
6. Patients who have received a live attenuated vaccine within 30 days prior to starting study treatment. Seasonal influenza vaccines that do not contain live viruses are permitted.
7. Patients who are currently participating in another clinical trial and receiving study treatment, or who have participated in a clinical trial and received investigational drug or device treatment within 4 weeks prior to enrollment.
8. Patients who have received any anti-tumor therapeutic agents containing traditional Chinese medicine ingredients within 4 weeks prior to starting study treatment.
9. Patients who have previously received an allogeneic tissue/organ transplant.
10. Patients who are expected to require any other form of anti-tumor therapy during the course of the study.
11. Patients who are receiving radiotherapy, with the exception of: 1) local radiotherapy for brain lesions, refer to exclusion criterion 25; 2) palliative radiation for bone metastases, provided that it is completed at least 7 days prior to randomization and the patient's condition is stable.
12. Patients with angina, myocardial infarction, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, unstable arrhythmia, pulmonary embolism, or treatment with percutaneous transluminal coronary angioplasty or coronary artery bypass grafting within 6 months prior to study treatment.
13. Patients with hypertension (defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg) or CTCAE Grade ≥2 hypotension.
14. Patients with uncontrolled or symptomatic hypercalcaemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN).
15. Patients with known history of or current hearing injury or Grade ≥2 peripheral neuropathy as defined by CTCAE v5.0 criteria (only for patients treated with cisplatin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization to the date of first documented disease progression (assessed by a blinded independent central review [BICR] according to RECIST v1.1) or death from any cause, whichever occurs first,assessed up to 6months.

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Beijing Chest Hospital, Beijing
  - Binzhou Medical University Hospital, Binzhou
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing University Three Gorges Hospital, Chongqing
  - Harbin Medical University Cancer Hospital, Ha’erbin
  - Anhui Provincial Cancer Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Jiangmen Central Hospital, Jiangmen
  - Yunan Cancer Hospital, Kunming
  - Linyi People's Hospital, Linyi
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Guangxi Medical University Cancer Hospital, Nanning
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - The Second People's Hospital of Neijiang, Neijiang
  - Shanghai Chest Hospital, Shanghai
  - First Hospital of Shanxi Medical University, Taiyuan
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Second People's Hospital of Yibin, Yibin
  - General Hospital of Ningxia Medical University, Yinchuan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhoukou Central Hospital, Zhoukou